CLINICAL TRIAL: NCT00989469
Title: SORAFENIB (NEXAVAR®) in Combination With Irinotecan in the Second Line Treatment or More of Metastatic Colorectal Cancer With K-RAS Mutation : a Multicentre Two-part Phase I/II Study.
Brief Title: Sorafenib With Irinotecan in Metastatic Colorectal Cancer (mCRC) and K-RAS Mutation
Acronym: NEXIRI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEXIRI
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sorafenib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib and irinotecan (Experimental)
  Interventions: Drug: Nexavar (Sorafenib) and irinotecan (Campto)

INTERVENTIONS:
Drug: Nexavar (Sorafenib) and irinotecan (Campto) — Sorafenib administrated continuously orally 400 mg twice daily (a daily total dose of 800 mg). Irinotecan 180 mg/m² will be administered IV for 90 minutes every 2 weeks. The first dose of sorafenib will be administered after the first perfusion of irinotecan 180 mg/m² at the first infusion

SUMMARY:
A multicentre two-part phase I/II study evaluating response and safety of SORAFENIB in combination with irinotecan in the second line treatment or more of metastatic colorectal cancer with K-RAS mutation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Written informed consent
* Histologically proven adenocarcinoma of the colon or rectum asymptomatic primary tumour or surgically removed mCRC patients with previously unresectable metastatic disease
* Patient with at least one tumoral lesion: measurable in a unidimensional way with a spiral scanner according to RECIST, no previous irradiation in this area
* Disease progression after irinotecan-based chemotherapy
* Disease progression after one or more previous lines of chemotherapy received in metastatic situation
* WHO <= 2
* Patient having a mutated KRAS on 12 or 13 codons on the primary tumour or a metastasis
* Adequate liver function : Bilirubin ≤ 1,5 x UNL, ASAT ou ALAT ≤ 2,5 x UNL (or < 5 x UNL for subjects having a hepatic insufficiency in connection with hepatic metastases)
* Polynuclear neutrophils ≥ 1 500/mm3
* Haemoglobin > 10g/dl
* Platelets ≥ 100 000/mm3
* Amylase and lipase < 1,5 x UNL
* Serum Creatinin < 1,5 x UNL
* Adapted contraceptive measures during treatment and continued at least three months after end of the treatment
* Life expectancy > 3 months
* Affiliated to or benefiting from health insurance

Exclusion Criteria:

* Gilbert's disease
* Brain metastases or carcinomatous symptomatic meningitis
* Exclusive bone metastasis
* Previous cancers not considered as cured in the 5 years before inclusion (except for baso-cellular skin carcinoma) Surgery (except diagnostic biopsy) or radiotherapy within 4 weeks before inclusion
* Disorders of the cardiac rhythm requiring an anti-asynchronous treatment (except beta blockers or digoxine within the framework of a chronic auricular fibrillation), unstable coronaropathy or myocardial infarction < 6 months, congestive cardiac failure > Rank II NYHA (Grade 2), uncontrolled arterial hypertension
* Previous epilepsy crises requiring long term antiepileptic treatment Previous organ transplant requiring immunosuppressor treatment Severe bacterial or fungus infection (> Grade 2 NCI CTC version 3) Known HIV Infection
* Long term treatment by known inductors of the CYP 3A4 like Rifampicin, Millepertuis (hypericum perforatum), Phenytoin, Carbamazepin, Phenobarbital, Dexamethasone et Ketonazole
* Known allergy to one of the therapeutic agents
* Reasons (psychological, family, social or geographical) that could compromise the participation of the patient in the study
* Intestinal malabsorption or gastro-intestinal surgery being able to affect Sorafenib absorption. Occlusive or sub-occlusive syndrome.
* Dysphagic patient or patient not being able to take treatment by orally inflammatory
* Chronic digestive disease involving chronic diarrhoea (NCI N+Bethesda >= 1.2g)
* Participation in another clinical trial within 30 days before the start of this study
* Other concomitant experimental drugs or other concomitant anticancer agents (except Irinotecan and Sorafenib)
* Medical or psychological state that in the opinion of the investigator will not allow the patient to terminate the study or to understand and sign the informed consent form
* Pregnancy and breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
disease control | 6 months

SECONDARY OUTCOMES:
Assessment of adverse events by using the NCI-CTCAE version 3 scale | 6 months
progression free survival | 24 months
overall survival | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmannuelle SAMALIN-SCALZI, Dr, Principal Investigator — CRLC Val d'Aurelle-Paul Lamarque
Locations (5):
- France (5):
  - Centre Oscar Lambret, Lille
  - Hopital Saint Eloi, Montpellier
  - Centre Rene Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Robert Debre, Reims

REFERENCES:
- [Result] Samalin E, Bouche O, Thezenas S, Francois E, Adenis A, Bennouna J, Taieb J, Desseigne F, Seitz JF, Conroy T, Galais MP, Assenat E, Crapez E, Poujol S, Bibeau F, Boissiere F, Laurent-Puig P, Ychou M, Mazard T. Sorafenib and irinotecan (NEXIRI) as second- or later-line treatment for patients with metastatic colorectal cancer and KRAS-mutated tumours: a multicentre Phase I/II trial. Br J Cancer. 2014 Mar 4;110(5):1148-54. doi: 10.1038/bjc.2013.813. Epub 2014 Jan 9. PMID 24407191